CLINICAL TRIAL: NCT07253844
Title: Effects of Transverse Abdominis Activation and Rectus Abdominis Strengthening on Inter-rectus Distance and Core Stability Among Patients With Diastasis Rectus Abdominis
Brief Title: Effects of Transverse Abdominis Activation and Rectus Abdominis Strengthening on Inter-rectus Distance and Core Stability
Acronym: TrA RA IRD DRA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/025
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Diastasis Recti Abdominis (DRA)
Keywords: Diastasis Rectus Abdominus; Inter rectus distance; Rectus abdominus strenghtheing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, blinding of participants and therapists was not be feasible. However, to minimize assessment bias, outcome assessors remained blinded to group allocations which establishing a single-blind study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Transverse abdominis activation) (Experimental)
  Interventions: Other: Transverse Abdominis activation exercises
- Group B (Rectus abdominis strengthening) (Experimental)
  Interventions: Other: Rectus Abdominis Strengthening exercises
- Group C (Transverse abdominis activation +rectus abdominis strengthening) (Experimental)
  Interventions: Other: combined protocol of both transverse abdominis activation and rectus abdominis strengthening.

INTERVENTIONS:
Other: Transverse Abdominis activation exercises — Group A (TAA) will perform abdominal drawing-in maneuvers (ADIM) in crook lying, side lying, and quadruped positions. They will be instructed to gently draw the belly button inward toward the spine without moving the pelvis or rib cage, emphasizing breathing coordination and pelvic floor co-activation. In the supervised phase, participants will perform 3 sets of 10 repetitions, with each contraction held for 10-20 seconds, and a rest interval of 3 minutes between sets
  Arms: Group A (Transverse abdominis activation)
Other: Rectus Abdominis Strengthening exercises — Group B (RAS) will perform exercises in supine lying with knees bent, including partial curl-ups, reverse crunches, pelvic tilts, and leg raises with abdominal bracing. The command will be tighten your abdominals as if bracing for a punch, and lift without straining your neck. Each supervised session will include 3 sets of 10-15 repetitions per exercise, progressing in difficulty using added resistance if tolerated, with a 3-minute rest interval between sets
  Arms: Group B (Rectus abdominis strengthening)
Other: combined protocol of both transverse abdominis activation and rectus abdominis strengthening. — Group C (TAA+RAS) will perform a hybrid protocol integrating both TrA activation and RA strengthening exercises. Each session will begin with ADIM in crook lying, side lying, and quadruped positions, followed by RA exercises including curl-ups, pelvic tilts, and leg raises. The command will be to activate your deep core with breathing, then strengthen your outer abdominals through controlled movements. Each supervised session will consist of 3 sets of 10 repetitions for TrA exercises (10-20 seconds hold) and 3 sets of 10-15 repetitions for RA exercises, with a rest period of 3 minutes between all sets.
  Arms: Group C (Transverse abdominis activation +rectus abdominis strengthening)

SUMMARY:
This randomized controlled trial aims to compare the effects of Transverse Abdominis (TrA) activation, Rectus Abdominis (RA) strengthening, and their combined approach on inter-rectus distance (IRD) and core stability in postpartum women diagnosed with diastasis rectus abdominis (DRA). Thirty-three participants will be randomly allocated into three groups and will complete a six-week exercise program at the Pakistan Society for the Rehabilitation of the Disabled (PSRD) Hospital, Lahore. The study will use real-time ultrasound and pressure biofeedback assessment to evaluate changes in IRD and core stability. It is hypothesized that TrA activation and the combined intervention will produce greater improvements compared to RA strengthening alone.

DETAILED DESCRIPTION:
Background and Rationale:

Diastasis Rectus Abdominis (DRA) is a prevalent postpartum musculoskeletal condition characterized by the separation of the rectus abdominis muscles along the linea alba, resulting in impaired trunk stability, abdominal weakness, and postural dysfunction. Despite its high prevalence, DRA remains underdiagnosed and undertreated, particularly in developing countries where structured rehabilitation protocols are lacking. Physiotherapy-based interventions focusing on abdominal muscle retraining and core stability have been shown to improve outcomes; however, the relative effectiveness of Transverse Abdominis (TrA) activation, Rectus Abdominis (RA) strengthening, and their combined approach remains uncertain.

Objectives:

This randomized controlled trial aims to compare the effects of TrA activation, RA strengthening, and their combination on inter-rectus distance (IRD) and core stability among postpartum women with DRA.

Methods:

This three-arm, parallel-group randomized controlled trial will be conducted at the Pakistan Society for the Rehabilitation of the Disabled (PSRD) Hospital, Lahore, Pakistan. A total of 33 postpartum women aged 20-40 years, diagnosed with DRA (6 months to 2 years postpartum), will be recruited using non-probability convenience sampling. Participants will be randomly assigned into three groups (n = 11 per group):

Group A (TAA): Transverse Abdominis Activation exercises

Group B (RAS): Rectus Abdominis Strengthening exercises

Group C (TAA + RAS): Combined TrA activation and RA strengthening protocol

Each participant will undergo a 6-week intervention program, including three supervised sessions per week for 3 weeks, followed by a 3-week home exercise program. Each session will last 30-45 minutes and will be supervised by a licensed physical therapist at PSRD.

Outcome Measures:

Primary Outcome: Change in Inter-Rectus Distance (IRD), measured via real-time ultrasound imaging (7.5 MHz linear probe) at three anatomical sites (4.5 cm above, at, and 4.5 cm below the umbilicus), pre- and post-intervention.

Secondary Outcome: Core stability, assessed using a Pressure Biofeedback Unit (PBU) during the abdominal drawing-in maneuver (ADIM) in crook-lying position. Participants will aim to reduce pressure by 6-10 mmHg from a 40 mmHg baseline and sustain the contraction for 10 seconds; the mean of three trials will be recorded.

Randomization and Blinding:

Participants will be randomized using Randomized Allocation Software (Version 1.0) in a 1:1:1 ratio. Due to the exercise-based nature of the interventions, blinding of participants and therapists is not feasible; however, the outcome assessor will remain blinded to group assignments, ensuring a single-blind design.

Data Analysis:

Statistical analysis will be performed using SPSS version 26. Data will first be tested for normality using the Shapiro-Wilk test. A two-way mixed ANOVA will be applied to assess both within-subject effects (time: pre vs. post) and between-subject effects (group: TAA, RAS, TAA+RAS), as well as the interaction effect (time × group) on IRD and core stability outcomes. Post-hoc pairwise comparisons with Bonferroni correction will identify specific between-group differences. Statistical significance will be set at p < 0.05 with a 95% confidence interval.

Expected Clinical Significance:

It is hypothesized that TrA activation exercises will lead to a greater reduction in IRD and improvement in core stability compared to RA strengthening alone. The combined exercise group (TAA + RAS) is expected to demonstrate the most comprehensive benefits due to synergistic activation of both deep and superficial abdominal muscles. The study outcomes are anticipated to provide evidence-based guidance for physiotherapists in postpartum rehabilitation, contributing to the development of standardized, non-invasive exercise protocols for DRA management and improved quality of life in postpartum women.

ELIGIBILITY:
Inclusion Criteria:

. Postpartum women diagnosed with DRA

* Multigravida
* Delivered a singleton pregnancy via vaginal breech or instrumental delivery

Exclusion Criteria:

. Pregnancy

* Abdominal and pelvic hernias or severe musculoskeletal conditions
* Patients with abdominal and pelvic surgery
* Patients with disc herniation

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 33 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Inter-rectus Distance (IRD) | Baseline: Before starting the intervention Post-intervention: At the end of 6 weeks of the exercise program
  The Inter-rectus Distance (IRD) is the measurement of the separation between the two rectus abdominis muscles along the linea alba. It is assessed using ultrasound imaging while the participant is in a supine position with knees bent.. A high-frequency (7.5 MHz) linear probe will be placed on the abdomen while the patient lies on their back. Images will be taken at three points above, at, and below the belly button.

SECONDARY OUTCOMES:
Core stability | Baseline (pre-intervention) and 6 weeks (post-intervention)
  core stability was assessed using the pressure biofeedback unit (PBU), a reliable and non-invasive tool designed to evaluate the activation and control of deep abdominal muscles, particularly TrA. The PBU consists of a pressure cuff connected to an analog pressure gauge and provides visual feedback on pressure changes in response to subtle lumbo pelvic movements (57). For assessment, participants were positioned in a crook lying position, and the cuff was positioned under the lumbar spine (L4-L5 region). The device was inflated to a baseline pressure of 40 mmHg, and participants will be instructed to perform the abdominal drawing-in maneuver, aiming to reduce the pressure by 6-10 mmHg without moving the pelvis or spine. They were asked to maintain this contraction for 10 seconds, and the procedure will be repeated three times, with the average score recorded for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad tariq Shafi, BSPT,tDPT, Study Chair — Lahore University of Biological and Applied Sciences
Locations (2):
- Pakistan (2):
  - Lahore University of biological and applied sciences, Lahore, Punjab Province
  - Pakistan Society for Rehabilitation of Differently Abled, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including demographic characteristics (age, parity, BMI), baseline and post-intervention ultrasound measurements of inter-rectus distance (IRD), abdominal muscle strength scores, and functional outcome or patient-reported measures related to abdominal function. Data will also include group allocation (Transverse Abdominis Activation or Rectus Abdominis Strengthening) for analysis comparison. All shared data will be stripped of any personal identifiers to ensure participant confidentiality. The shared dataset will be available in a coded format for secondary analysis and research transparency purposes only.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The de-identified individual participant data (IPD) and supporting documents (study protocol, statistical analysis plan, and informed consent form) will be made available after completion of data analysis and publication of the main study results, approximately 6 months after study completion. The data will remain accessible for a period of 3 years following the publication date. Requests for data access must be submitted to the principal investigator and will be reviewed to ensure appropriate use consistent with ethical and confidentiality standards. No personally identifiable information will be shared at any stage.
Access Criteria: De-identified individual participant data (IPD) and supporting information (study protocol, analysis plan, and informed consent form) will be available to qualified researchers, academicians, and postgraduate students conducting studies related to abdominal rehabilitation, physiotherapy, or maternal health. Access will be provided upon reasonable written request to the principal investigator, accompanied by a brief research proposal and data use agreement ensuring confidentiality. Approved users will receive the data in an electronic, password-protected format via institutional email. The data will be shared solely for academic and non-commercial research purposes, with strict adherence to ethical and privacy standards.

REFERENCES:
- [Background] Benjamin DR, Frawley HC, Shields N, van de Water ATM, Taylor NF. Relationship between diastasis of the rectus abdominis muscle (DRAM) and musculoskeletal dysfunctions, pain and quality of life: a systematic review. Physiotherapy. 2019 Mar;105(1):24-34. doi: 10.1016/j.physio.2018.07.002. Epub 2018 Jul 24. PMID 30217494
- [Background] Olsson A, Woxnerud K, Kiwanuka O, Sandblom G, Stackelberg O. The TOR concept (training, operation, and rehabilitation) applied to a cohort of postpartum women with training-resistant symptomatic rectus diastasis: evaluation 1 year after surgery. BJS Open. 2023 Jan 6;7(1):zrac162. doi: 10.1093/bjsopen/zrac162. PMID 36734959
- [Background] Gluppe SL, Hilde G, Tennfjord MK, Engh ME, Bo K. Effect of a Postpartum Training Program on the Prevalence of Diastasis Recti Abdominis in Postpartum Primiparous Women: A Randomized Controlled Trial. Phys Ther. 2018 Apr 1;98(4):260-268. doi: 10.1093/ptj/pzy008. PMID 29351646
- [Background] Pascoal AG, Dionisio S, Cordeiro F, Mota P. Inter-rectus distance in postpartum women can be reduced by isometric contraction of the abdominal muscles: a preliminary case-control study. Physiotherapy. 2014 Dec;100(4):344-8. doi: 10.1016/j.physio.2013.11.006. Epub 2014 Jan 18. PMID 24559692
- [Background] Berg-Poppe P, Hauer M, Jones C, Munger M, Wethor C. Use of exercise in the management of postpartum diastasis recti: a systematic review. The Journal of Women's & Pelvic Health Physical Therapy. 2022;46(1):35-47.